CLINICAL TRIAL: NCT05992051
Title: Effects of Online Exercise Intervention on Physical and Mental Conditions in Young Adults With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Principal Investigator, JINGHUA QIAN, Professor, deputy dean of School of Sports Medicine and Rehabilitation, Beijing Sport University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20212069
Record Dates: First submitted 2023-07-29; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Chronic Non-specific Neck Pain
Keywords: chronic neck pain; non-specific neck pain
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with 39 adults with self-reported chronic neck pain recruited. They were randomly assigned into two groups. The experimental group received online exercise therapy and the control group received conventional exercise therapy.
  Participants in both groups completed the same exercise program three times a week for six weeks. Visual analogue scale (VAS), the Neck Disability Index (NDI), Work Limitations Questionnaire (WLQ) and The Hospital Anxiety and Depression Scale (HADS) and its subscales were evaluated. Participants were assessed at baseline and at 6 weeks while the changes in WLQ were assessed biweekly. To ensure the effectiveness of online exercise therapy, therapists delivered the online exercise 3 times a week for 6 weeks, with videoconferencing once a week and posting of exercise record on social media twice a week.
Who Masked: Outcomes Assessor
Masking Description: This experiment was performed as a single-blind experiment. The outcomes assessors are specialized personnel who do not participate in the trial intervention process and are not clear about the grouping of participants situation and the intervention situation. Outcome statistics were also performed by dedicated data analysts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- online exercise therapy (Experimental): The participants had weekly online exercise meetings with the physiotherapist in a group of 3-5 participants using online meeting app. Then the participants performed the remaining two sessions of exercises themselves weekly. All the participants of the experimental group received a package of exercise pamphlet and a video disc containing 17-minute exercise demonstrations by the physiotherapist.
  At baseline, the suitable elastic bands (Thera-band®) for performing the exercises were selected by testing the 15 repetitions maximum (15RM) of the Modified Brügger's Exercise (MBE) and the Modified Proprioceptive Neuromuscular Facilitation Diagonal Flexion Exercise (MPNFDFE) for the participants of both the experimental group and control group.
  Participants performed the following exercises three times a week for six weeks at home:
  A. Warm-up exercises B. Cranio-cervical flexion exercises C. Strength-endurance exercises D. Scapular stabilization exercises E. Stretching exercises
  Interventions: Behavioral: Exercise Therapy
- conventional exercise therapy (Active Comparator): Participants in the control group completed the same exercise program three times a week for six weeks with face-to-face mode delivery by physiotherapists.
  At baseline, the suitable elastic bands (Thera-band®) for performing the exercises were selected by testing the 15 repetitions maximum (15RM) of the Modified Brügger's Exercise (MBE) and the Modified Proprioceptive Neuromuscular Facilitation Diagonal Flexion Exercise (MPNFDFE) for the participants of both the experimental group and control group.
  Participants performed the following exercises three times a week for six weeks in a group of 3-5 participants in the laboratory of the Sport Medicine and Rehabilitation School of the Beijing Sport University:
  A. Warm-up exercises B. Cranio-cervical flexion exercises C. Strength-endurance exercises D. Scapular stabilization exercises E. Stretching exercises
  Interventions: Behavioral: Exercise Therapy

INTERVENTIONS:
Behavioral: Exercise Therapy — Exercise therapy is considered as the integral component of interventions for chronic non-specific neck pain. It includes different type resistance training, range of motion exercises and stretching exercises to improve neck condition and release symptoms.

SUMMARY:
This study aimed to compare the efficacy of online exercise therapy with conventional exercise therapy on pain, function, psychological status and work efficiency of young adults with chronic neck pain. A randomized clinical trial recruiting 39 university students with self-reported chronic neck pain was conducted. Participants were randomly assigned into the experimental group receiving online exercise therapy and the active control group receiving conventional exercise therapy. Participants in both groups completed the same exercise program 3 sessions per week for 6 weeks, with either face-to-face or online mode of delivery by physiotherapists. The pain level was assessed using visual analogue scale (VAS) based on average and at maximum intensity. Neck function and work limitations were assessed by the Neck Disability Index (NDI) and Work Limitations Questionnaire (WLQ) respectively. The Hospital Anxiety and Depression Scale (HADS) and its subscales (HADS-A and HADS-D) were used to evaluate the overall symptoms, levels of anxiety and depression respectively. Participants were assessed at baseline and at 6 weeks while the changes in WLQ were assessed biweekly.

It is hypothesized that, young adults with chronic neck pain, both the online and conventional exercise interventions could improve their pain level, neck disability, anxiety state and work efficiency, and the online exercise intervention appeared feasible as an alternative treatment option for them.

DETAILED DESCRIPTION:
Study Title： Effects of Online Exercise Intervention on Physical and Mental Conditions in Young Adults with Chronic Neck Pain Study Population： The target participants were adults with self-reported non-specific neck pain for more than three months. They were recruited through posters and social media in the campus of the Beijing Sport University.

Study Design： The present study was an assessor blinded randomized controlled trial conducted according to the Declaration of Helsinki (World Medical Association, 2013). The Institutional Review Board of the Beijing Sport University approved the study (reference number: 2023006H). A randomized clinical trial recruiting 39 university students with self-reported chronic neck pain was conducted. Participants were randomly assigned into the experimental group receiving online exercise therapy and the active control group receiving conventional exercise therapy. Participants in both groups completed the same exercise program 3 sessions per week for 6 weeks, with either face-to-face or online mode of delivery by physiotherapists.

Sample Size Assessment： The sample size for the study was calculated to be 32 using the G*Power 3.1.9.2 (University Kiel, Germany), with an estimated effect size of group difference of 0.9 in primary outcomes and a level of significance of 0.05, statistical power of 80% with 2-tailed independent sample t test. With an anticipated dropout rate of 15%, a total of 39 participants was required.

Study Duration： Totally 8 weeks, including 1-week baseline testing, 6-week intervention and 1-week post intervention testing.

Study Intervention Description： Participants in both groups completed the same exercise program three times a week for six weeks with either face-to-face or online mode of delivery by physiotherapists.

Primary Objective： The primary objective is to study the effectiveness of online and conventional exercise therapy on pain level and function in adults with chronic neck pain. There were three primary outcomes, including average and maximum neck pain using visual analog scale (VAS), and Neck Disability Index (NDI).

Secondary Objectives： The secondary objectives are investigating the effectiveness of online and conventional exercise therapy on mental condition and working efficacy in adults with chronic neck pain. There were two secondary outcomes: anxiety and depression measured with the Hospital Anxiety and Depression Scale (HADS) and work efficiency assessed with the Work Limitations Questionnaire (WLQ).

Statistical analysis: Continuous data were expressed as means and standard deviations. Categorical data were shown as frequencies or percentages, with group comparisons performed using the Fisher exact test. The normality of continuous data was checked with the Shapiro-Wilk test. The change scores of the primary and secondary outcome variables from baseline to end of intervention between the 2 groups were compared using independent sample t test with approximate data normality. The Cohen's effect sizes of between-group comparisons were calculated. The Mann-Whitney U test was used for group comparison of non-normal continuous data. Within-group comparisons were done using paired sample t test.

ELIGIBILITY:
Inclusion Criteria:

* adults between 18 and 50 years of age with neck pain (from occiput to 7th cervical vertebra) for at least 3 months
* a score of >= 4/50 on the Neck Disability Index.

Exclusion Criteria:

* adults with a history of previous neck surgery, cervical radiculopathy, acute neck injury or fracture
* persons who had more than two hours of moderate intensity exercise or more than four hours of low intensity exercise in a week
* persons who had received any form of physiotherapy treatment in the last 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
visual analog scale (VAS) | measured at baseline prior to randomization and after the 6-week intervention period
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. In this study, the VAS is used to measure the average and maximum neck pain level. The outcome is measured with 100-mm visual analog scale (VAS), in which 0 indicating no pain and 10.0 indicating unbearable pain.
Neck Disability Index (NDI) | measured at baseline prior to randomization and after the 6-week intervention period
  The Neck Disability Index (NDI) is a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain. The NDI consists of 10 items related to pain intensity, headache, concentration and different physical activities. The score of each item ranges from 0 to 5. The maximum total score is 50 and the final score will be standardized into 0 to 100. The higher the score of the NDI, the more severe the neck dysfunction is.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | measured at baseline prior to randomization and after the 6-week intervention period
  The Hospital Anxiety and Depression Scale (HADS) was devised 30 years ago by Zigmond and Snaith to measure anxiety and depression in a general medical population of patients. In this study, it was used to measure the mental condition of participants. The scale comprises 14 questions which related 2 underlying sub-scale dimensions, anxiety (HADS-A) and depression (HADS-D) respectively. Each subscale has 7 items and each item is scored with 0-3 points. The minimum and maximum values of the HADS are 0 and 42. The higher the score, the more severe the condition is. The minimum and maximum values of the subscales are 0 and 21, and higher scores mean a worse outcome. Those with score ≥8 on HADS-A or HADS-D were considered to be at high risk of having anxiety or depression.
Work Limitations Questionnaire (WLQ) | measured at baseline prior to randomization and after the 2-week, 4-week, 6-week intervention period
  The Work Limitations Questionnaire (WLQ-25) is a 25-item objective measure used to evaluate at-work disability and productivity loss. It is a self-reported tool to evaluate the degree of difficulty in completing 25 specific tasks in the past 2 weeks. The score of each task ranges from 1 (no difficulty) to 5 (always having difficulties). The minimum and maximum values of the WLQ are 25 and 125. The higher the score, the lower the work efficiency is.

CONTACTS AND LOCATIONS:
Overall Officials: Jinghua Qian, Doctor, Study Chair — Beijing Sport University
Locations (1):
- School of Sports Medicine and Rehabilitation, Beijing Sport University, Beijing, Beijing Municipality, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT05992051/Prot_SAP_000.pdf